CLINICAL TRIAL: NCT05002621
Title: Exploratory Investigation of Changes in Gene Transcription and Immunophenotypes Following Mepolizumab Treatment for Asthma
Brief Title: Changes in Gene Transcription and Immunophenotypes Following Mepolizumab Treatment for Asthma
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Thanai Pongdee, Principal Investigator, Mayo Clinic
Other Study IDs: 20-005018
Record Dates: First submitted 2021-08-09; First posted 2021-08-12 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Eosinophilic Asthma
MeSH Terms: conditions — Pulmonary Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify gene transcripts after initiation of mepolizumab in individuals with severe eosinophilic asthma (SEA), and to determine the composition of immune cells present in the microenvironment of individuals with SEA after initiation of mepolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Diagnosis of SEA by a health care provider
* History of an absolute eosinophil count ≥ 300/mm^3
* Prescription for mepolizumab provided during course of routine clinical care but mepolizumab not yet started

Exclusion Criteria:

* Age < 18 years old.
* Pregnancy.
* Currently using or have used within 3 months of the initial baseline visit any biologic or immunomodulatory therapy with the exception of #3.
* Currently using or any prior use of rituximab.
* History of upper/lower respiratory tract infection or asthma exacerbation within the previous four weeks of the first baseline visit.
* Any prior history of malignancy, autoimmune disease, or immune deficiency.
* Any other significant medical issue as determined by the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve twenty adult (≥18yo) individuals with a diagnosis of severe eosinophilic asthma (SEA) who have been prescribed mepolizumab during their course of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Expressed gene transcripts | Baseline and 4, 8, and 12 weeks post-initiation of mepolizumab
  RNA sequencing will be performed from collected peripheral blood mononuclear cells (PBMCs) at four time points to compare changes in expressed gene transcripts.
Composition of immune cell subsets | Baseline and 4, 8, and 12 weeks post-initiation of mepolizumab
  CyTOF mass cytometry (50 test immune phenotype panel including cell surface markers, transcription factors, and cytokines) will be performed on PBMCs isolated from peripheral blood at four time points.

CONTACTS AND LOCATIONS:
Overall Officials: Thanai Pongdee, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials